CLINICAL TRIAL: NCT04028219
Title: Transgender In Transition: Metabolism, Behaviour and Psychopathology in Transsexual Patients Following Hormonal Treatment
Brief Title: Transgender In Transition
Acronym: TRANSIT
Status: Recruiting | Type: Observational
Sponsor: Universitätsklinikum Hamburg-Eppendorf (Other)
Responsible Party: Sponsor
Other Study IDs: TRANSIT
Record Dates: First submitted 2019-07-14; First posted 2019-07-22 (Actual); Last update posted 2022-11-08 (Actual); Status verified 2022-11

CONDITIONS: Gender Incongruence
MeSH Terms: conditions — Gender Dysphoria

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Transgender patients: Gender dysphoric patients undergoing hormone treatment
  Interventions: Diagnostic Test: Online surveys

INTERVENTIONS:
Diagnostic Test: Online surveys — Psychometric measures within 14 online surveys, which is one at each assessment point (before and 3, 6, 9, 12, 24, 36, 48, 60, 72, 84, 96, 108, 120 months after hormonal therapy).

SUMMARY:
Prospective trial in gender dysphoric patients who undergo gender-affirming hormone therapy, aiming to investigate psychological, biological and behavioural consequences of hormonal therapy.

DETAILED DESCRIPTION:
Gender-affirming hormone treatment impacts myriads of body functions, from which it has to be assumed that only a minority has already been elucidated so far. This project aims to investigate the consequences and health-related outcomes of various hormone therapies in the treatment of gender dysphoric patients. The main scientific interest lies in the research of the effects of sex hormones on psychological, metabolic and behavioural parameters. For this purpose, various investigations are aimed at, including a clinical-diagnostic interview (external rating) and psychometric measurements in self-rating, behavioral experiments (e.g. in a virtual reality Elevated Plus Maze and the computer-based Ultimatum Game) and genetic investigation of the body's own materials (blood samples, stool samples, hair samples and saliva samples). The results of this study should form the basis to better understand consequences of the long-term administration of sex hormones.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of gender incongruence (ICD-11) or gender dysphoria (DSM-5)
* written informed consent following adequate oral and written Information
* before gender-affirming hormonal treatment

Exclusion Criteria:

* pregnancy or breast-feeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Individuals with gender incongruence undergoing gender-affirming hormone treatment
Sampling Method: Non-Probability Sample
Enrollment: 750 (Estimated)
Dates: Start 2019-05-15 (Actual); Primary Completion 2024-05-15 (Estimated); Study Completion 2034-05-15 (Estimated)

PRIMARY OUTCOMES:
Mini International Neuropsychiatric Interview (MINI; Lecrubier et al., 1997) | 10 years
  The Mini International Neuropsychiatric Interview (MINI; Lecrubier et al., 1997) is a short structured clinical interview which enables researchers to make diagnoses of psychiatric disorders according to DSM-IV or ICD-10 and was designed for epidemiological studies and multicenter clinical trials.

SECONDARY OUTCOMES:
Alcohol Use Disorders Identification Test-Consumption (Audit C; Wade et al., 2014) | 10 years
  The Alcohol Use Disorders Identification Test-Consumption (Audit C; Wade et al., 2014) measures the consumption of alcohol in the past 12 months via a self-rating of 3 items. For the planned study, further equivalent versions for the consumption of nicotine and cannabis were adapted with 9 items covering consumption behaviour.
Transgender Congruence Scale (TCS; Kozee et al., 2012) | 10 years
  The Transgender Congruence Scale (TCS; Kozee et al., 2012) measures gender congruence via self-rating through twelve items and two subscales (congruence with appearance & acceptance of gender identity) within the past two weeks.
Gender Congruence and Life Satisfaction Scale (GCLS; Jones et al., 2018) | 10 years
  The Gender Congruence and Life Satisfaction Scale (GCLS; Jones et al., 2018) measures gender congruence and life satisfaction via self-rating through 38 items and seven subscales (genitals, breast, other secondary sexual characteristics, recognition of gender role, physical and emotional intimacy, physiological function and life satisfaction) with a time frame of six months.
Brief Symptom Inventory (BSI; Derogatis and Melisaratos, 1983) | 10 years
  The Brief Symptom Inventory (BSI; Derogatis and Melisaratos, 1983) measures psychiatric symptoms via self-rating with a total of 53 items in the areas of somatisation, compulsivity, insecurity in social contact, depression, anxiety, aggression, phobic fear, paranoid thinking and psychoticism. The inventory refers to a description of the symptoms within the past week.
Short Form 36 (SF-36; Jenkinson et al., 1993) | 10 years
  The Short Form 36 (SF-36; Jenkinson et al., 1993) measures the health-related quality of life in the past month via self-rating with a total of 36 items, whereby it refers to the following areas: Vitality, physical functioning, physical pain, general health perception, physical role function, emotional role function, social functioning and psychological well-being.
Patient Health Questionnaire-9 (PHQ-9; Löwe et al., 2004) | 10 years
  The Patient Health Questionnaire-9 (PHQ-9; Löwe et al., 2004) measures the severity of depression symptoms via self-rating. The PHQ-9 is one of the most widely used depression questionnaires worldwide and enables the estimation of realistic basic rates of diagnosis of major depression.
Beck Scale for Suicidal Ideation (BSSI; Beck et al., 1979) | 10 years
  The Beck Scale for Suicidal Ideation (BSSI; Beck et al., 1979) measures the degree of suicidal tendencies within the past week by self-rating with 21 items.
Questionnaire for the Evaluation of Psychotherapy Processes / Fragebogen zur Evaluation von Psychotherapieverläufen (FEP-2; Lutz et al., 2009) | 10 years
  The questionnaire for the evaluation of psychotherapy processes (FEP-2; Lutz et al., 2009) is a self-rating instrument comprising 40 items and is used for quality assurance in psychiatric/psychotherapeutic treatments. This questionnaire covers the areas of well-being, symptom burden, interpersonal problems and incongruity within the past week.
Barratt Impulsivity Scale / Barratt Impulsivitäts Skala (BIS-15; Meule et al., 2011) | 10 years
  The short form of the Barratt Impulsivity Scale (BIS-15; Meule et al., 2011) measures various forms of impulsivity (motor, planning, attention) via self-rating based on 15 items.
Questionnaire for Empathy and Changing Perspectives / Fragebogen für Empathie und Perspektivenübernahme (EP; Paulus, 2009) | 10 years
  The Questionnaire for Empathy and Changing Perspectives (EP; Paulus, 2009) uses self-rating with a total of 18 items to determine the ability to empathize and to change perspectives in the areas of empathy, social sensitivity and prosocial behaviour.
Autism-Spektrum-Quotient (AQ-10; Sappok et al., 2015) | 10 years
  The short version of the autism spectrum quotient (AQ-10; Sappok et al., 2015) is a screening instrument for recording autistic traits via self-rating that comprises 10 items.
Rosenberg Self-Esteem Scale (RSES; Robins et al., 2001) | 10 years
  The Rosenberg Self-Esteem Scale (RSES; Robins et al., 2001) measures self-esteem via self-rating with 10 items.
Internalized Stigma of Mental Illness Inventory (ISMI-9; Hammer and Toland, 2017) | 10 years
  The Internalized Stigma of Mental Illness Inventory (ISMI-9; Hammer and Toland, 2017) measures the tendency towards self-stigmatization in psychiatric populations via self-rating with 9 items.
Multidimensional Sexuality Questionnaire (MSQ; Snell et al., 1993) | 10 years
  The Multidimensional Sexuality Questionnaire (MSQ; Snell et al., 1993) is a self-rating instrument for recording various psychological dimensions of sexuality. For economic reasons, a selection of three subscales (sexual anxiety, depression and satisfaction) will be specified in the current project. This selection comprises a total of 14 items.
Sexual Desire Inventory (SDI; Spector et al., 1996) | 10 years
  The Sexual Desire Inventory (SDI; Spector et al., 1996) measures sexual desire in the past month via self-rating with 13 items. There are two different subscales for desire with and desire without social interaction (solitary and dyadic sexual desire).
Side Effects of Hormonetherapy Inventory / Fragebogen zu Nebenwirkungen der Hormontherapie | 10 years
  This specially for the current study developed questionnaire on side effects of hormone therapy uses self-rating to record various psychological and physiological symptoms that were observed during transition treatments with gender, sexual desire and sexual desire in 23 items.
Borderline Symptom List (BSL-23; Bohus et al., 2009) | 10 years
  The Borderline Symptom List (BSL-23; Bohus et al., 2009) measures symptoms that typically occur in the context of borderline personality disorder via self-rating with 34 items. The time frame refers to the previous week.
Core Autogynephilia Scale (CAS; Blanchard, 1989) | 10 years
  The Core Autogynephilia Scale (CAS; Blanchard, 1989) meassures autogynephile tendencies via self-rating with 9 items. For the planned study, an equivalent version (Core Autoandrophilia Scale) was adapted to be able to measure autoandrophilic tendencies equally.
OPD Structure Questionnaire Short Version / OPD Strukturfragebogen Kurzversion (OPD-SFK; Ehrenthal et al., 2015) | 10 years
  The OPD Structure Questionnaire Short Version (OPD-SFK; Ehrenthal et al., 2015) uses self-rating with a total of 12 items in order to measure structural abilities in the dimensions of self-perception, contact design and relationship model.
Personality Inventory for DSM-5 Brief Form / Persönlichkeitsinventar für DSM-5 (PID-5-BF; Anderson et al., 2016) | 10 years
  The personality inventory for DSM-5 Brief Form (PID-5 BF; Anderson et al., 2016) measures pathological personality traits via self-rating with a total of 25 items, which are described by the following subscales: Negative affectivity, closure, antagonism, disinhibition and psychoticism.
Childhood Trauma Questionnaire (CTQ; Bernstein et al., 2003) | 10 years
  The Childhood Trauma Questionnaire (CTQ; Bernstein et al., 2003) is a self-evaluation tool suitable for retrospectively recording abuse and neglect in childhood and adolescence. The CTQ measures more than traumatic events in the narrower sense (according to DSM-IV and ICD-10). The CTQ scales include abuse (with three subscales: emotional, physical, sexual) and neglect (with two subscales: emotional and physical). The subscales consist of five items each. In addition, a further scale (three items) is provided to measure tendencies to trivialize or deny child abuse experiences. The items are rated on a 5-level scale (1-5 from 'not at all' to 'very often').
ENRICHD Social Support Inventory (ESSI; Mitchell et al., 2003) | 10 years
  The ENRICHD Social Support Inventory (ESSI; Mitchell et al., 2003) measures the perception of social support via self-rating with 5 items.
Perseverative Thinking Questionnaire (PTQ; Ehring et al., 2011) | 10 years
  The Perseverative Thinking Questionnaire (PTQ; Ehring et al., 2011) measures the extent of brooding thoughts via self-rating with 15 items.
2 Subscales of the Sensation Seeking Scale-V (SSS-V; Zuckerman, 2007): thrill- and adventure seeking & experience-seeking | 10 years
  The Sensation Seeking Scale-V (SSS-V; Zuckerman, 2007) measures individual differences in sensation seeking via self-rating on the basis of various dimensions, which are: Thrill and Adventure Seeking (TAS), Disinhibition (Dis), Experience Seeking (ES), and Boredom Susceptibility (BS). Each subscale contains 10 items. For economic reasons, only two subscales (TAS & ES) are used in the current project.
Acrophobia Questionnaire (AQ; Cohen, 1977) | 10 years
  The Acrophobia Questionnaire (AQ; Cohen, 1977) is a self-rating questionnaire measuring acrophobia (fear of heights). The AQ describes 20 situations (e.g. standing next to an open window in an upper floor), which are often regarded by acrophobic patients as anxiety provoking and asks the extent of the anxiety (0-6) and avoidance behaviour (0-3). A total of 0-180 points can be achieved.
Trust and Reciprocity Questionnaire (TR; Cox, 2004) | 10 years
  The Trust and Reciprocity Questionnaire (TR; Cox, 2004) measures trust and reciprocity via self-rating with 9 items.
Client Satisfaction Questionnaire (CTQ-8) / Fragebogen zur Patientenzufriedenheit (ZUF-8; Schmidt et al., 2002) | 10 years
  The Client Satisfaction Questionnaire CSQ-8 (ZUF-8; Schmidt et al., 2002) is a validated self-rating questionnaire on satisfaction with treatment in psychiatric clinics. This questionnaire has been adapted for the current study so that patient satisfaction with hormone treatment is measured.

CONTACTS AND LOCATIONS:
Overall Officials: Johannes Fuß, MD, Principal Investigator — Institute for Sex Research, Sexual Medicine and Forensic Psychiatry
Locations (5):
- Germany (3):
  - Universitätsklinikum Frankfurt, Frankfurt am Main, Hesse
  - University Medical Center Hamburg-Eppendorf, Hamburg
  - Medical Center of the Ludwig-Maximilians-University of Munich, Munich
- Switzerland (2):
  - Universitätsspital Basel, Basel
  - UniversitätsSpital Zürich, Zurich

IPD SHARING:
Plan to Share IPD: Undecided